CLINICAL TRIAL: NCT04612738
Title: Project Talk Trial: Engaging Underserved Communities in End-of-life Conversations: a Cluster, Randomized Controlled Trial
Brief Title: Project Talk Trial: Engaging Underserved Communities in End-of-life Conversations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Hospice Foundation of America (Unknown); University of Kentucky (Other)
Responsible Party: Principal Investigator, Lauren Van Scoy, Associate Professor of Medicine, Humanities, and Public Health Sciences; Co-director of Penn State Mixed Methods Core, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00014689
Record Dates: First submitted 2020-10-12; First posted 2020-11-03 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-05

CONDITIONS: Advance Care Planning; Advance Directives; Terminal Illness; Chronic Illness; Communication
Keywords: serious games
MeSH Terms: conditions — Chronic Disease; Communication

STUDY DESIGN:
Intervention Model Description: This is a 3-armed, cluster randomized controlled trial that will compare the efficacy of two evidenced based interventions, with a nationally-promoted structured workbook, Conversation Project (CP) Starter Kit; and use of a Placebo/Attention control, non-ACP game called Table Topics. The primary outcome is completion of an advance directive 6 months post-intervention.
Who Masked: Investigator
Masking Description: The principal investigator and statistical teams will be blinded to the allocation of study participants to the study arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1:Advance care planning conversation game, 'Hello' (Active Comparator): The 'Hello' game is a commercially available serious game that consists of 32 questions prompting players to share their values, goals, and beliefs about end-of-life issues. The game is played with 4 - 5 players, with each receiving a game booklet and chips. A play reads the first question in the book. Then each player writes down their answers individually and takes turns sharing their answers with the group. Players control what they share, how long they share and when to move to the next questions. During the conversation, plays can acknowledge others for a thoughtful, poignant or even funny comments by giving them a chip. A pre-game coin flip determines whether the player with the most chips wins the game (heads) or player with the least chips win (tails) the game.
  Other names; previously name "My Gift of Grace"
  Interventions: Behavioral: Hello (serious game)
- Group 2: The Conversation Project (CP) Starter Kit (Active Comparator): The 'CP Starter Kit' (available for free online) is an 11-page workbook with open- ended prompts to consider one's values and preferences for end-of-life care, who to talk with about one's wishes, and suggestions on how to do so.
  Interventions: Behavioral: The Conversation Project (CP) Starter Kit
- Group 3: Control Arm (Placebo control game, 'Table Topics') (Placebo Comparator): A placebo/attention control l conversation game called 'Table Topics' will be used. Table Topics is a general conversation starter game that is unrelated to advance care planning. It involves answering open-ended questions in a group setting about a variety of topics.
  Interventions: Other: Table Topics (general conversation game)

INTERVENTIONS:
Behavioral: Hello (serious game) — Commercially available, 'Hello' 32 is a serious game that consists of 32 questions prompting players to share their values, goals, and beliefs about end-of-life issues. The creators developed the questions following interviews with palliative care clinicians, hospice nurses, and funeral directors, and then revised them through a series focus groups with >100 patients/caregivers from diverse backgrounds.
  Arms: Group 1:Advance care planning conversation game, 'Hello'
Behavioral: The Conversation Project (CP) Starter Kit — The CP Starter Kit is one of the most widely promoted and disseminated ACP tools nationwide, is available for free online, and does not require a healthcare professional for use. Like 'Hello', it is intended to help individuals have end-of-life conversations with loved ones. The 11-page workbook has open- ended prompts to consider one's values and preferences for end-of-life care, who to talk with about one's wishes, and suggestions on how to do so. It also prompts participants to rank priorities on a 5-point scale (e.g., What are your concerns about treatment? 1= I'm worried I won't get enough care, 5= I'm worried I'll get overly aggressive care). The CP website provides resources for running a community event using the 'CP Starter Kit', including a 23-page manual, "Coaching the Conversation- A Guide to Facilitating Conversation Groups," with details on hosting a community-based program.
  Arms: Group 2: The Conversation Project (CP) Starter Kit
Other: Table Topics (general conversation game) — Table topics is a popular, commercially available conversation starter game that consists of question cards to prompt conversations (e.g., 'What do you love about your hometown?').
  Arms: Group 3: Control Arm (Placebo control game, 'Table Topics')

SUMMARY:
Compared to the general population, individuals from underserved communities are more likely to receive low quality end-of-life care and unwanted, costly and burdensome treatments due in part to a lack of advance care planning (ACP; the process of discussing wishes for end-of-life care with loved ones/clinicians and documenting them in advance directives).

This study will use existing, trusted, and respected social networks to evaluate two conversation-based tools intended to engage underserved individuals in discussions about end-of-life issue and motivate them to carry out ACP behaviors.

Through this study, investigators will learn how best to engage underserved populations in ACP so as to: 1) increase the likelihood that patients from underserved communities will receive high-quality end-of-life care; 2) address health disparities related to end-of-life treatments; and 3) reduce unnecessary suffering for patients and their families.

DETAILED DESCRIPTION:
The overall project goal of this 3-armed cluster, randomized control trial in underserved, diverse communities is to determine whether playing a serious conversation game called Hello is more effective than other advance care planning (ACP) approaches, or usual care (i.e., simply distributing an advance directive [AD]). The investigators will randomize 75 underserved communities across the US. The primary outcome is completion of a visually verified AD; secondary outcomes include performance of other ACP behaviors.

Many Black/African Americans and Latina/Latino patients are more likely to receive low quality end-of- life medical care than White individuals- in fact, they are 3 times more likely than white Americans to die after a lengthy intensive care unit stay. Advance care planning (ACP)- the process of discussing one's wishes with loved ones and clinicians, and then documenting them in an advance directive (AD)- can help reduce these health inequities by preventing costly/burdensome treatments that are unlikely to reduce suffering or improve quality of life. Though ~60% of Americans engage in ACP, <25% of underserved populations have done so- in large part due to distrust of the healthcare system/clinicians, and reluctance to discuss death and dying.

This study leverages underserved communities' existing, trusted social networks to deploy two community-based ACP interventions and study their mechanisms of action. By identifying which interventions increase engagement in ACP in underserved communities (and why), this project will help improve quality of end-of-life care, reduce unnecessary suffering, and end-of-life healthcare costs which conserves public health resources.

ELIGIBILITY:
Inclusion Criteria Community Hosts

1. Ability to recruit 20 individuals from underserved populations to attend a community event
2. Experience hosting a community event
3. Experience working with underserved populations
4. Participation in a series of mandatory live study-related web-based trainings
5. Completes a research site agreement

Research Participants

1. Adults over the age of 18 years old in underserved populations
2. Able to speak and read English and/or Spanish
3. Have not completed an AD within the previous 5 years
4. All participants regardless of health status
5. Individuals from the same household can enroll

Exclusion Criteria Community Hosts

1. Inability to recruit 20 individuals from underserved populations
2. Inexperience for hosting a community event
3. Inexperience working with underserved populations
4. Unable to attend a series of mandatory live study-related web-based trainings
5. Do not provide informed consent
6. Do not complete a research site agreement
7. Previously hosted a Hello project event

Research Participants

1. Anyone <18 years of age
2. Anyone not able to speak and read English and/or Spanish
3. Have significant difficulties with hearing or speaking difficulties by self-report
4. Completed an AD in the past 5 years
5. Do not provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2022-03-19 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Rates of Completion of a Visually Verified Advance Directive | 6 months post-intervention
  Study team confirms completion of a signed advance directive

SECONDARY OUTCOMES:
Rates of Other Advance Care Planning (ACP) behaviors | 6 months post-intervention
  Performance of other ACP behaviors such as self-reported ACP completion, discussions with loved ones, financial preparations
Advance Care Planning Engagement Survey | Baseline (Day 0); 6 months post-intervention
  This short-version survey measures readiness to perform ACP

OTHER OUTCOMES:
Previous Exposure to ACP Interventions and Advance Directives | Baseline (Day 0)
  This baseline assessment of ACP completion and exposure
Healthcare System Distrust Scale | Baseline (Day 0)
  An assessment of two primary domains of distrust (values and competence) in the healthcare system. This is a 9-item measure, scored 9 - 45 with 9 being the least amount of distrust.
Experience and Comfort with Games Questionnaire | Baseline (Day 0 )
  This is a 4-item questionnaire to control for whether participants with familiarity with games respond differently to the intervention.
Acceptability of Intervention Measure | Immediately post-intervention (Day 0)
  This 3-item measure to access a participants' perceived acceptability of the intervention
Conversation Satisfaction Questionnaire | Immediately post-intervention (Day 0)
  This is a 8-item questionnaire that assesses a participant's satisfaction with conversation, with each item scored on a 1 - 7 scale, with 1 being lowest conversation satisfaction. The items are averaged for the final score ranging 1 - 7 with 7 indicating the highest conversation satisfaction.
Communication Quality Analysis (CQA) Measure | post-intervention
  This is a validated coding method which measures communication quality using outside observer ratings of audio recordings of an intervention.
Qualitative Community Host Interview | 2 weeks post-intervention
  A follow-up qualitative telephone interview will explore implementation and process outcomes.
Participant Follow-up Qualitative Telephone Interview | 2 weeks post-intervention
  A qualitative follow-up interview with a subset of intervention participants to explore experiences and perceptions of the intervention, adverse events and cultural norms related to healthcare and advance care planning.
Six-Month Participant Follow-up Telephone Interview | 6 months post-intervention
  This follow-up phone interview includes questionnaires that access whether participants went on to perform various behaviors related to advance care planning, as well as explore qualitatively how sociocultural environment impacts the advance care planning experience.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren J. Van Scoy, MD, Principal Investigator — Penn State Milton S. Hershey Medical Center; Penn State University College of Medicine
Locations (80):
- United States (80):
  - Pincham-Lincoln Community Center, Athens, Alabama
  - Kingman Regional Medical Center, Kingman, Arizona
  - Accord Health Group, Show Low, Arizona
  - El Rio Neighborhood Center, Tucson, Arizona
  - Promotores y Promotoras, Santa Paula, California
  - Our Lady of Solitude, Soledad, California
  - Vitas, Walnut Creek, California
  - University of Colorado Hospital, Aurora, Colorado
  - HopeWest Montrose, Montrose, Colorado
  - Stamford Senior Center, Stamford, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - DeSoto Memorial Hospital, Arcadia, Florida
  - High Point Neighborhood Family Center, Clearwater, Florida
  - St. Phillip AME Church, Tallahassee, Florida
  - City of Temple Terrace, Omar K. Lightfoot Center, Temple Terrace, Florida
  - 47Million Reasons Healthcare Movement, West Palm Beach, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Helene S. Mills, Atlanta, Georgia
  - Seniors First of GA, Atlanta, Georgia
  - Gilmer County Senior Center, Ellijay, Georgia
  - Colquitt Regional Medical Center, Moultrie, Georgia
  - University of Chicago Medical Ctr, Chicago, Illinois
  - St. Thomas the Apostle Catholic Church, Crystal Lake, Illinois
  - Lightways Hospice & Serious Illness Care, Joilet, Illinois
  - First Baptist Church, Quincy, Illinois
  - Trinity Lutheran Church, Cherokee, Iowa
  - Hospice & Home Care of Reno, Hutchinson, Kansas
  - Center for Practical Bioethics, Lawrence, Kansas
  - Ohio County Senior Centers, Hartford, Kentucky
  - Bluegrass Care Navigators, Lexington, Kentucky
  - United Crescent Hill Ministries, Louisville, Kentucky
  - Union County Senior Services, Morganfield, Kentucky
  - Hospice of Lake Cumberland, Somerset, Kentucky
  - Acadian Advocacy Network, Lafayette, Louisiana
  - St. Mary's Health System, Lewiston, Maine
  - East End Community Center, Portland, Maine
  - Good Hope Union UMC, Silver Spring, Maryland
  - Holy Cross Health, Silver Spring, Maryland
  - Grove Hall Senior Center, Boston, Massachusetts
  - Community Economic Development Center, New Bedford, Massachusetts
  - Christ Temple Church, Muskegon Heights, Michigan
  - Northeast Mississippi Coalition Against COVID-19, Belden, Mississippi
  - Elder Law Project of North Mississippi Rural Legal Services, Oxford, Mississippi
  - Columbia Senior Activity Center, Columbia, Missouri
  - Patch Center, St Louis, Missouri
  - Washoe Tribe Health Center, Gardnerville, Nevada
  - Reformed Church of Freehold, Freehold, New Jersey
  - Booker T. Washington CES, Las Cruces, New Mexico
  - Corsi Senior Center, New York, New York
  - Hospice of St. Lawrence Valley, Potsdam, New York
  - University of Rochester Medical Center, Rochester, New York
  - Greater Vision United Methodist Church, Huntersville, North Carolina
  - Plaza on Princess, Wilmington, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Cleveland Clinic, Akron, Ohio
  - Hospice of the Western Reserve, Cleveland, Ohio
  - McGregor Gardens, Cleveland, Ohio
  - Hope Behavioral Health, Cleveland, Ohio
  - Eastside Fellowship Ministries, Columbus, Ohio
  - Hospice Care of Middletown, Middletown, Ohio
  - Hospital Council of Northwest Ohio, Toledo, Ohio
  - Harney County Home Health & Hospice, Burns, Oregon
  - Stuart Community Center, Carlisle, Pennsylvania
  - Villa Schiano, Elizabethville, Pennsylvania
  - Latino Hispanic American Community Center, Harrisburg, Pennsylvania
  - People's Community Baptist Church, Harrisburg, Pennsylvania
  - Hospice and Community Care, Lancaster, Pennsylvania
  - St. Mark Missionary Baptist Church, Bennettsville, South Carolina
  - Welcome Home of Chattanooga, Chattanooga, Tennessee
  - All Saints Episcopal Church, Cameron, Texas
  - Turner Alumni Association, Carthage, Texas
  - Dorothea Street Community Center, Crane, Texas
  - Como Community Center, Fort Worth, Texas
  - Georgetown Public Library, Georgetown, Texas
  - Choice Hospice, Sulphur Springs, Texas
  - Sunshine Terrace Foundation, Logan, Utah
  - Luray Fire Department, Luray, Virginia
  - Carmel Baptist Church, Winchester, Virginia
  - Grayland Hall, Grayland, Washington
  - Ocean Beach Hospital, Ilwaco, Washington

IPD SHARING:
Plan to Share IPD: No
Our study team is highly motivated to share data with outside investigators as a means to ensure reproducibility of findings, further the scientific inquiry, and to avoid unintentional duplication of research. However, only de-identified data would be shared from this database under the auspices of the PI, and only after securing a Data Transfer Agreement. Whether the individual participant data or aggregated data will be determined based on each individual request.

REFERENCES:
- [Derived] Costigan HJ, VanDyke E, Calo WA, Tucci A, Van Scoy LJ; Project Talk Trial Collaborative Working Group Members. Adapting Advance Care Planning Interventions for Hispanic Communities Across the U.S. Am J Hosp Palliat Care. 2025 Dec;42(12):1290-1297. doi: 10.1177/10499091241306427. Epub 2024 Dec 19. PMID 39700514
- [Derived] Van Scoy LJ, Levi BH, Bramble C, Calo W, Chinchilli VM, Currin L, Grant D, Hollenbeak C, Katsaros M, Marlin S, Scott AM, Tucci A, VanDyke E, Wasserman E, Witt P, Green MJ. Comparing two advance care planning conversation activities to motivate advance directive completion in underserved communities across the USA: The Project Talk Trial study protocol for a cluster, randomized controlled trial. Trials. 2022 Sep 30;23(1):829. doi: 10.1186/s13063-022-06746-3. PMID 36180899

DOCUMENTS (4):
  • Informed Consent Form: Project Talk Trial-ICF-Hello-10122020 (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT04612738/ICF_001.pdf
  • Informed Consent Form: Project Talk Trial-ICF-Hosts-10122020 (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT04612738/ICF_003.pdf
  • Informed Consent Form: Project Talk Trial-ICF-CPKit-10102020 (2020-10-10): https://cdn.clinicaltrials.gov/large-docs/38/NCT04612738/ICF_002.pdf
  • Informed Consent Form: Project Talk Trial-ICF-Control-10122020 (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT04612738/ICF_000.pdf